CLINICAL TRIAL: NCT07358169
Title: The Impact of Mirror Therapy on Motor Recovery and Pain of Hemiparetic Arm Post Stroke: A Randomized Controlled Trial
Brief Title: Mirror Therapy on Motor Recovery and Pain of Hemiparetic Arm
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant Prof, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mirror therapy
Record Dates: First submitted 2026-01-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Stroke (CVA) or TIA; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Other): usual hospitl care
  Interventions: Other: Control
- mirror group (Experimental)
  Interventions: Other: technique; Other: Control

INTERVENTIONS:
Other: technique — the participant performs arm exercise behind mirror
  Arms: mirror group
Other: Control — the control group receive usual hospital care

SUMMARY:
evaluate the effect of mirror therapy on motor recovery and pain of hemiparetic arm post stroke

ELIGIBILITY:
Inclusion Criteria:

* First stroke attack (ischemic and haemorrhagic )
* Unilateral stroke with hemiparesis
* Able to understand simple verbal language

Exclusion Criteria:

* Severe cognitive impairments.
* Orthopedic or rheumatologic problems restricting upper extremity motor function.
* Contraindications to mirror therapy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Motor Function Assessment | 3 weeks
  measured by Fugl-Meyer Assessment for upper limb motor function. to describe impairment severity, quantify motor recovery, guide treatment planning, and evaluate outcomes. The scale comprises five domains with a maximum total score of 226 points (Motor 100; Sensation 24; Balance 14; Joint ROM 44; Joint Pain 44).
  Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
  Points are divided among the domains as follows:
  Motor score: ranges from 0 (hemiplegia) to 100 points (normal motor performance). Divided into 66 points for upper extremity and 34 points for the lower extremity.
  Sensation: ranges from 0 to 24 points. Divided into 8 points for light touch and 16 points for position sense.
  Balance: ranges from 0 to 14 points. Divided into 6 points for sitting and 8 points for standing.

SECONDARY OUTCOMES:
Functional independence | 3 weeks
  Functional independence (measured by Modified Rankin Scale). it is a 7-point scale (0-6) that measures disability after a stroke or neurological event, assessing the ability to perform daily activities, from no disability (0) to death (6).
  The Modified Rankin Scale Grade mRS 0 No symptoms at all
  1. No significant disability: despite symptoms, able to carry out all usual duties and activities
  2. Slight disability: unable to perform all previous activities but able to look after own affairs without assistance
  3. Moderate disability: requiring some help but able to walk without assistance
  4. Moderately severe disability: unable to walk without assistance and attend to own bodily needs without assistance
  5. Severe disability: bedridden, incontinence, and requiring constant nursing care and attention
  6. Death
Pain assessment | 3 weeks
  Pain assessment (measured by Numeric Pain Rating Scale.) it is a 11-point scale (0-10) where patients rate their pain intensity, with 0 meaning no pain and 10 representing the worst imaginable pain.
  scoring system 0: No Pain 1-3: Mild Pain 4-6: Moderate Pain 7-10: Severe Pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Mansoura, Egypt